CLINICAL TRIAL: NCT04792840
Title: Lymphedema and Skeletal Events in Older Patients Receiving Adjuvant Hormonal and Radiotherarpy in Breast Cancer
Brief Title: Skeletal Events of Hormonal Treatment and Radiotherapy in Patient With Breast Cacer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed gamal hussein, residant doctor, Assiut University
Other Study IDs: events in breast cancer
Record Dates: First submitted 2020-11-25; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Femara Pill — study effect on bone
  Other Names: radiothearpy

SUMMARY:
study of lymphedema and skeletal events in breast cacer patient receiving adjuvant hormonal therapy and radiothearpy

DETAILED DESCRIPTION:
In the United States, it is estimated that there are more than 3.8 million living women has a history of invasive breast cancer, and 268,600 women will be newly diagnosed in 2019. Sixty-four percent of breast cancer survivors (more than 2.4 million women) are ≥ 65 years, whereas 7% are aged younger than 50 years 1.

The most common treatment of early stage (stage I or II) breast cancer is breast-conserving surgery (BCS) with adjuvant radiation therapy (49%) and 34% of patients undergo mastectomy. In contrary, more than two-thirds (68%) of patients with stage III disease undergo mastectomy and most of them receive adjuvant chemotherapy 2.

Some of the most debilitating morbidity after surgery and radiotherapy for breast cancer is related to treatment of the axilla. This includes persistent arm lymphoedema, impaired shoulder mobility and brachial plexopathy. Other exogenous factors have an influence on the risk of radiotherapy-related morbidity as patients' age and obesity 3.

Lymphedema of the arm occurs in 19.9% of women who undergo axillary lymph node dissection and in 5.6% of women who have a sentinel lymph node biopsy 4. Irradiation of the regional lymph nodes may increase the risk, especially among patients receiving axillary lymph node dissection 5.

Early diagnosis of lymphedema is important for optimizing its treatment and preventing its progression 6. Some forms of cancer rehabilitation may reduce the risk and lessen the severity of this condition 7, 8.

Treatment with adjuvant aromatase inhibitors (AI), which is generally reserved for postmenopausal women, can cause osteoporosis 9.

Osteoporosis, a process of bone mineral density (BMD) reduction, is accelerated by estrogen deficiency in postmeno¬pausal women. Tamoxifen reduces BMD in premenopausal women, while promotes bone formation in postmenopausal patients. On the other hand, adjuvant aromatase inhibitors (AIs) therapy enhances the BMD decrease to about 2.5% per year, due to a long lasting significant deprivation of circula¬tory and tissue estrogens 10. In the bone companion study of the MA.17 trial, patients treated with anastrozole reported a significant decreases in BMD (~4%), compared to those treated with tamoxifen 11.

Dual energies' X ray absorptiometry (DXA) scan is the current validated 'gold standard' for the diagnosis of osteoporosis, fracture risk estimation and follow up of anti osteoporotic treatment 12-14, since it is non invasive, simple, precise, fast, less expensive than other imaging techniques, including computed tomography and magnetic resonance imaging, and more sensitive than quantitative ultrasound (QUS) 15.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal patients with positive diagnosis of stage 1-3 breast cancer and planned AI (anastrazole, letrozole) adjuvant treatment will be included in the study.
* Patients without known osteoporosis will included in the study, and before AI treatment began.
* Conventional RT course must be completed (50 Gy/25 fractions, 2 Gy/fraction, 5 days/week).
* Patients continue to receive adjuvant hormonal treatment (aromatase inhibitors) or adjuvant target therapy (trastuzumab) while monitoring late toxicities

Exclusion Criteria:

* Male patients
* Metastatic disease at presentation
* No definitive surgery
* Carcinoma in situ or other rare tumors of the breast as phyllodes tumors.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: older patient with breat cancer who receives hormonal treatment and radiothearpy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Skeletal events caused by hermonal treatment | basline
  Hermonal treatment in breast Cancer patients may caused osteoporosis that can be measured by dexascan
Radiotherapy and arm edema | Baseline
  Radiothearpy on axilla my increase arm edema in breast cancer patients measuredvby arm circumference in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: hanan g. mostafa, prof dr, Study Director — Assiut University; mohammed a. mohmmed, dr, Study Director — Assiut University; maha s. el naggar, dr, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided